CLINICAL TRIAL: NCT04640337
Title: Influence of Placebo on Intratissue Percutaneous Electrolysis (IPE) Treatment in Patients With Patellar Tendinopathy
Brief Title: Influence of Placebo on Intratissue Percutaneous Electrolysis in Patellar Tendinopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Mercè Balasch i Bernat, Principal investigator, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1264955
Record Dates: First submitted 2020-11-10; First posted 2020-11-23 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Patellar Tendinopathy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants don't know to which intervention group they belong to. The outcomes assessor doesn't know to which intervention group the patient belongs to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group E1: IPE applied, participants believe they are receiving IPE. (Experimental): IPE will be applied following the standard protocol for PT. Participants will believe they are receiving IPE.
  Interventions: Other: IPE applied, participants believe they are receiving IPE
- Group E2: IPE applied, participants believe they are receiving placebo. (Placebo Comparator): IPE will be applied following the standard protocol for PT. Subjects will be led to believe that the intensity of the current is below the threshold necessary to cause changes in the tissue.
  Interventions: Other: IPE applied, participants believe they are receiving placebo
- Group P1: IPE not applied, participants believe they are receiving IPE. (Placebo Comparator): The needle will be inserted under the skin but the current will not be passing through. The subjects will see a shame video on the ultrasound screen so they will believe that the IPE is being performed.
  Interventions: Other: IPE not applied, participants believe they are receiving IPE
- Group P2: IPE not applied, participants believe they are receiving placebo. (Placebo Comparator): The needle will be inserted under the skin, subjects will be led to believe that the intensity of the current is below the threshold necessary to cause changes in the tissue.
  Interventions: Other: IPE not applied, participants believe they are receiving placebo

INTERVENTIONS:
Other: IPE applied, participants believe they are receiving IPE — Participants will receive a total of 3 sessions of IPE, with a time interval of one week between the 1st and 2nd session and 2 weeks between the 2nd and 3rd session. IPE will be applied following the standard protocol for PT. Participants will believe they are receiving IPE.
  Arms: Group E1: IPE applied, participants believe they are receiving IPE.
Other: IPE applied, participants believe they are receiving placebo — Participants will receive a total of 3 sessions of IPE, with a time interval of one week between the 1st and 2nd session and 2 weeks between the 2nd and 3rd session. IPE will be applied following the standard protocol for PT. Subjects will be led to belie
  Arms: Group E2: IPE applied, participants believe they are receiving placebo.
Other: IPE not applied, participants believe they are receiving IPE — Participants will receive a total of 3 sessions of IPE-placebo, with a time interval of one week between the 1st and 2nd session and 2 weeks between the 2nd and 3rd session. The needle will be inserted under the skin but the current will not be passing th
  Arms: Group P1: IPE not applied, participants believe they are receiving IPE.
Other: IPE not applied, participants believe they are receiving placebo — Participants will receive a total of 3 sessions of IPE-placebo, with a time interval of one week between the 1st and 2nd session and 2 weeks between the 2nd and 3rd session. The needle will be inserted under the skin, subjects will be led to believe that the intensity of the current is below the threshold necessary to cause changes in the tissue.
  Arms: Group P2: IPE not applied, participants believe they are receiving placebo.

SUMMARY:
The main aim of this study is to verify the influence of placebo on the effectiveness of Intratissue Percutaneous Electrolysis (IPE) in patients suffering from with chronic patellar tendinopathy (PT).

The secondary aim is to investigate the possible influence of the IPE on pain perception and conditioned pain modulation (CPM) in patients with chronic PT.

DETAILED DESCRIPTION:
The aim of this study is to investigate the influence of placebo on the effectiveness of Intratissue Percutaneous Electrolysis (IPE) in patients with chronic PT. For this purpose a randomized clinical trial will be carried out, with a sample of patients diagnosed of chronic PT based on signs, symptoms and clinical examination. Subjects will be randomly allocated to four different groups: group E1, IPE will be applied, participants will believe they are receiving IPE; group E2, IPE will be applied, participants will believe they are receiving placebo; group P1, IPE will not be applied, participants will believe they are receiving IPE; and group P2, IPE will not be applied, participants will believe they are receiving placebo.

IPE treatment will consist of a total of 3 sessions, with a time interval of one week between the 1st and 2nd sessions and 2 weeks between the 2nd and 3rd sessions.

To evaluate the effect of intervention, the subjects will be assessed at baseline (V0), one week after the end of the intervention (V1) and 3 weeks after the intervention (V2).

In V0, sociodemographic (sex, age, profession, height, body mass index (BMI), sport activity, hours of sport per week) and clinical data (associated pathologies, affected lower limb, dominant lower limb, duration of symptoms) will be registered. In each assessment time information regarding BMI, sports activity, hours of sport per week and location of pain will be obtained. Moreover, in all assessments participants were evaluated for four physical performance tests, pain and functional scales, ultrasound examination, pressure pain thresholds, conditioned pain modulation, and expectations questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* presenting the following signs and symptoms of patellar tendinopathy: pain when jumping, landing, running o changing direction, pain at the inferior pole of the patella, Victorian Institute of Sport Assessment-Patella (VISA-P) score <80, symptoms duration of at least 3 months.

Exclusion Criteria:

* prior knee surgery
* patients having received local corticosteroids injection in the tendon within the preceding 6 months
* patients presenting any inflammatory disease, metabolic bone disease, type II diabetes, fibromyalgia, hypercholesterolemia, pregnancy or chemotherapy within the 3 months prior to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10-16 (Actual); Primary Completion 2023-12-20 (Estimated); Study Completion 2024-03-20 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Baseline
  Knee pain intensity reported by the patient will be assessed using a 100-mm visual analogue scale (VAS, 0-100, 0=minimum score, 100=maximum score). Higher values represent a better outcome (less pain).
Pain intensity | One week post-intervention
  Knee pain intensity reported by the patient will be assessed using a 100-mm visual analogue scale (VAS, 0-100, 0=minimum score, 100=maximum score). Higher values represent a better outcome (less pain).
Pain intensity | Three weeks post-intervention
  Knee pain intensity reported by the patient will be assessed using a 100-mm visual analogue scale (VAS, 0-100, 0=minimum score, 100=maximum score). Higher values represent a better outcome (less pain).
Patellar tendon function | Baseline
  Victorian Institute of Sport Assessment-Patellar Tendon (VISA-P, 0-100, 0=minimum score, 100=maximum score) will aso be used to evaluate function of the patellar tendon. A score between 80-100 points is considered as the optimal outcome.
Patellar tendon function | One week post-intervention
  Victorian Institute of Sport Assessment-Patellar Tendon (VISA-P, 0-100, 0=minimum score, 100=maximum score) will aso be used to evaluate function of the patellar tendon. A score between 80-100 points is considered as the optimal outcome.
Patellar tendon function | Three weeks post-intervention
  Victorian Institute of Sport Assessment-Patellar Tendon (VISA-P, 0-100, 0=minimum score, 100=maximum score) will aso be used to evaluate function of the patellar tendon. A score between 80-100 points is considered as the optimal outcome.
Physical performance of the knee | Baseline
  Physical performance of the knee will be assessed by the Single Leg Decline squat (SLDS), which consists of performing a squat with one leg on a decline board with an angle of 25º.
Physical performance of the knee | One week post-intervention
  Physical performance of the knee will be assessed by the Single Leg Decline squat (SLDS), which consists of performing a squat with one leg on a decline board with an angle of 25º.
Physical performance of the knee | Three weeks post-intervention
  Physical performance of the knee will be assessed by the Single Leg Decline squat (SLDS), which consists of performing a squat with one leg on a decline board with an angle of 25º.
Cross-sectional area (CSA) of the patellar tendon | Baseline
  CSA at rest, with a knee flexion of 20º, will be measured by ultrasonography.
Cross-sectional area (CSA) of the patellar tendon | One week post-intervention
  CSA at rest, with a knee flexion of 20º, will be measured by ultrasonography.
Cross-sectional area (CSA) of the patellar tendon | Three weeks post-intervention
  CSA at rest, with a knee flexion of 20º, will be measured by ultrasonography.
Presence of neovascularity of the patellar tendon | Baseline
  The presence (yes/no) of neovascularity of the patellar tendon will be measured by ultrasonography.
Presence of neovascularity of the patellar tendon | One week post-intervention
  The presence (yes/no) of neovascularity of the patellar tendon will be measured by ultrasonography.
Presence of neovascularity of the patellar tendon | Three weeks post-intervention
  The presence (yes/no) and amount (0=no vascularity, 1=low fow, 2=mild flow, 3=high flow) of neovascularity of the patellar tendon will be measured by ultrasonography.
Amount of neovascularity of the patellar tendon | Baseline
  The amount (0=no vascularity, 1=low fow, 2=mild flow, 3=high flow) of neovascularity of the patellar tendon will be measured by ultrasonography.
Amount of neovascularity of the patellar tendon | One week post-intervention
  The amount (0=no vascularity, 1=low fow, 2=mild flow, 3=high flow) of neovascularity of the patellar tendon will be measured by ultrasonography.
Amount of neovascularity of the patellar tendon | Three weeks post-intervention
  The amount (0=no vascularity, 1=low fow, 2=mild flow, 3=high flow) of neovascularity of the patellar tendon will be measured by ultrasonography.

SECONDARY OUTCOMES:
Pressure Pain Thresholds (PPT) | Baseline
  PPTs will be recorded using an electronic algometer at the ipsilateral (affected) patellar tendon, the contralateral patellar tendon and the ipsilateral upper trapezius. Higher values represent a better outcome.
Pressure Pain Thresholds (PPT) | One week post-intervention
  PPTs will be recorded using an electronic algometer at the ipsilateral (affected) patellar tendon, the contralateral patellar tendon and the ipsilateral upper trapezius. Higher values represent a better outcome.
Pressure Pain Thresholds (PPT) | Three weeks post-intervention
  PPTs will be recorded using an electronic algometer at the ipsilateral (affected) patellar tendon, the contralateral patellar tendon and the ipsilateral upper trapezius. Higher values represent a better outcome.
Conditioned pain modulation (CPM) | Baseline
  CPM will be tested using the upper extremity submaximal effort tourniquet test.
Conditioned pain modulation (CPM) | One week post-intervention
  CPM will be tested using the upper extremity submaximal effort tourniquet test.
Conditioned pain modulation (CPM) | Three weeks post-intervention
  CPM will be tested using the upper extremity submaximal effort tourniquet test.
Patients' expectations | Baseline
  Patients' expectations with the treatment will be registered using an add-hoc questionnaire consisting of 2 questions: "What do you think will be the intensity of your pain when this intervention takes effect?" (NPRS, 0-10, 10 severe pain, 0=no pain) and "Do you expect to have more pain, less pain or the same intensity of pain after treatment?" (more pain, less pain, same pain).
Self-perceived change with the treatment | One week post-intervention
  Participants' will rate the results/outcomes obtained with the treatment by the Global rating of change scale (GROC) ((-7)-(+7), -7= very great deal worse, +7= very great deal better).
Self-perceived change with the treatment | Three weeks post-intervention
  Participants' will rate the results/outcomes obtained with the treatment by the Global rating of change scale (GROC) ((-7)-(+7), -7= very great deal worse, +7= very great deal better).
Self-perceived pain after treatment | One week post-intervention
  Self-perceived pain after treatment will be assessed by the question "What do you think your pain is like now (after treatment): more pain, less pain or the same pain intensity compared to before treatment?" (more pain, less pain, same pain).
Self-perceived pain after treatment | Three weeks post-intervention
  Self-perceived pain after treatment will be assessed by the question "What do you think your pain is like now (after treatment): more pain, less pain or the same pain intensity compared to before treatment?" (more pain, less pain, same pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Mercè Balasch i Bernat, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No